CLINICAL TRIAL: NCT00881985
Title: Effect of Continuous Positive Airway Pressure for Treatment of Obstructive Sleep Apnea on Drug-resistant Hypertension : A Randomized Controlled Trial
Brief Title: Effect of Continuous Positive Airway Pressure for Treatment of Obstructive Sleep Apnea on Resistant Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Professor Ip Sau Man Mary, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 09-051
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Resistant Hypertension; Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; resistant hypertension; refractory hypertension; continuous positive airway pressure; blood pressure control
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension | interventions — Continuous Positive Airway Pressure

ARMS (2):
- continuous positive airway pressure (Active Comparator)
  Interventions: Device: continuous positive airway pressure
- observation (No Intervention)

INTERVENTIONS:
Device: continuous positive airway pressure — Use CPAP whenever sleep
  Other Names: CPAP
  Arms: continuous positive airway pressure

SUMMARY:
The objectives of this study are to investigate the effect of continuous positive airway pressure (CPAP) treatment on blood pressure control and vascular inflammation in subjects with resistant hypertension and moderate obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Resistant hypertension is defined as blood pressure that remains above goal in spite of concurrent use of 3 antihypertensive agents of different classes. Resistant hypertension is defined in order to identify patients who are at risk of having secondary causes of hypertension, and who may benefit from specific diagnostic and therapeutic applications. Despite the fact that OSA is listed as one of the causes of resistant HT , paucity of works has demonstrated the magnitude of problems of untreated OSA in subjects with resistant HT. There is so far two study demonstrating the beneficial effect of CPAP treatment in subjects with resistant HT, though both studies were flawed by not including the control group, no randomization and limited sample size. We aim at conducting a randomized controlled study to explore the beneficial effect of CPAP treatment in subjects with OSA and resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65
* known hypertension on ≧ 3 anti-hypertensive drugs
* Apnea-hypopnea index ≧15
* able to give informed written consent

Exclusion Criteria:

* moderate renal impairment (glomerular filtration rate <30 mL/min/m2 )
* endocrine/renal/cardiac causes of secondary HT
* congestive heart failure and clinically fluid overloaded
* On drugs that elevates BP e.g. NSAID, steroid
* Non-compliance to anti-hypertensive medications
* Unstable medical conditions such as unstable angina, recent myocardial infarction/stroke within 3 months
* Active inflammatory/infective conditions e.g. rheumatoid arthritis
* Excessive sleepiness that can be risky e.g. occupational driver, machine operator
* Modification/changes of anti-hypertensive regimen within 8 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-03; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
mean systolic blood pressure | 8 weeks

SECONDARY OUTCOMES:
mean arterial blood pressure | 8 weeks
mean diastolic blood pressure | 8 weeks
high sensitivity C-reactive protein | 8 weeks
cardiac injury marker | 8 weeks
oxidative stress marker | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary SM Ip, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China

REFERENCES:
- [Background] Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, D'Agostino RB, Newman AB, Lebowitz MD, Pickering TG. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA. 2000 Apr 12;283(14):1829-36. doi: 10.1001/jama.283.14.1829. PMID 10770144
- [Background] Young T, Peppard P, Palta M, Hla KM, Finn L, Morgan B, Skatrud J. Population-based study of sleep-disordered breathing as a risk factor for hypertension. Arch Intern Med. 1997 Aug 11-25;157(15):1746-52. PMID 9250236
- [Background] Pepperell JC, Ramdassingh-Dow S, Crosthwaite N, Mullins R, Jenkinson C, Stradling JR, Davies RJ. Ambulatory blood pressure after therapeutic and subtherapeutic nasal continuous positive airway pressure for obstructive sleep apnoea: a randomised parallel trial. Lancet. 2002 Jan 19;359(9302):204-10. doi: 10.1016/S0140-6736(02)07445-7. PMID 11812555
- [Background] Becker HF, Jerrentrup A, Ploch T, Grote L, Penzel T, Sullivan CE, Peter JH. Effect of nasal continuous positive airway pressure treatment on blood pressure in patients with obstructive sleep apnea. Circulation. 2003 Jan 7;107(1):68-73. doi: 10.1161/01.cir.0000042706.47107.7a. PMID 12515745
- [Background] Norman D, Loredo JS, Nelesen RA, Ancoli-Israel S, Mills PJ, Ziegler MG, Dimsdale JE. Effects of continuous positive airway pressure versus supplemental oxygen on 24-hour ambulatory blood pressure. Hypertension. 2006 May;47(5):840-5. doi: 10.1161/01.HYP.0000217128.41284.78. Epub 2006 Apr 3. PMID 16585412
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM. Resistant hypertension: diagnosis, evaluation, and treatment. A scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Hypertension. 2008 Jun;51(6):1403-19. doi: 10.1161/HYPERTENSIONAHA.108.189141. Epub 2008 Apr 7. PMID 18391085
- [Background] Logan AG, Perlikowski SM, Mente A, Tisler A, Tkacova R, Niroumand M, Leung RS, Bradley TD. High prevalence of unrecognized sleep apnoea in drug-resistant hypertension. J Hypertens. 2001 Dec;19(12):2271-7. doi: 10.1097/00004872-200112000-00022. PMID 11725173
- [Background] Grote L, Hedner J, Peter JH. Sleep-related breathing disorder is an independent risk factor for uncontrolled hypertension. J Hypertens. 2000 Jun;18(6):679-85. doi: 10.1097/00004872-200018060-00004. PMID 10872551
- [Background] Lavie P, Hoffstein V. Sleep apnea syndrome: a possible contributing factor to resistant. Sleep. 2001 Sep 15;24(6):721-5. doi: 10.1093/sleep/24.6.721. PMID 11560187
- [Background] Logan AG, Tkacova R, Perlikowski SM, Leung RS, Tisler A, Floras JS, Bradley TD. Refractory hypertension and sleep apnoea: effect of CPAP on blood pressure and baroreflex. Eur Respir J. 2003 Feb;21(2):241-7. doi: 10.1183/09031936.03.00035402. PMID 12608436
- [Background] Martinez-Garcia MA, Gomez-Aldaravi R, Soler-Cataluna JJ, Martinez TG, Bernacer-Alpera B, Roman-Sanchez P. Positive effect of CPAP treatment on the control of difficult-to-treat hypertension. Eur Respir J. 2007 May;29(5):951-7. doi: 10.1183/09031936.00048606. Epub 2007 Feb 14. PMID 17301092
- [Derived] Lui MM, Tse HF, Lam DC, Lau KK, Chan CW, Ip MS. Continuous positive airway pressure improves blood pressure and serum cardiovascular biomarkers in obstructive sleep apnoea and hypertension. Eur Respir J. 2021 Nov 4;58(5):2003687. doi: 10.1183/13993003.03687-2020. Print 2021 Oct. PMID 33795324